CLINICAL TRIAL: NCT04695184
Title: The Value of Subjective Near-infrared Fluorescence Guidance in Assessment of Perfusion During Restorative Ileal Pouch Formation and Ileal-pouch-anal Anastomosis
Brief Title: Subjective Near-infrared Fluorescence Guidance in Perfusion Assessment of Ileal Pouch Formation and Ileal-pouch-anal Anastomosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benjamin Weixler, Attending Physician, Assistant Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA4/116/19/1
Record Dates: First submitted 2020-12-22; First posted 2021-01-05 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis; Colorectal Cancer; Crohn Disease; Familial Adenomatous Polyposis; Crohn Colitis; Ileal Pouch
Keywords: indocyanine green; restorative proctocolectomy; ileal pouch-anal anastomosis; subjective perfusion rate; near-infrared fluorescence; ulcerative colitis; anastomotic leak; pouchitis
MeSH Terms: conditions — Colitis, Ulcerative; Colorectal Neoplasms; Crohn Disease; Adenomatous Polyposis Coli; Anastomotic Leak; Pouchitis

STUDY DESIGN:
Intervention Model Description: This is a non randomised prospective cohort study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-NIRF Imaging (Other): ICG-NIRF imaging is used intraoperatively to visualise precisely the blood supply and bowel perfusion rate in the area of ileal pouch formation and the ileal pouch-anal anastomosis.
  Interventions: Diagnostic Test: ICG-NIRF Imaging

INTERVENTIONS:
Diagnostic Test: ICG-NIRF Imaging — intraoperative NIRF Imaging using the fluorescence agent ICG (indocyanine-green) at regions of interest before (T1) + after pouch construction (T2) + after ileoanal anastomosis (T3)

SUMMARY:
In this prospective, non-randomized cohort study, real-time intraoperative visualization using near-infrared-fluorescence by indocyanine green injection (ICG-NIRF) is performed at three time points during ileal pouch reconstruction. The intraoperative imaging findings are then analysed and correlated with the 30 day postoperative clinical outcome including occurrence of anastomotic leak of the pouch.

DETAILED DESCRIPTION:
Near-infrared-fluorescence by indocyanine green (ICG-NIRF) utilises the fluorescent property of intravenously injected indocyanine green (ICG) as an intravascular indicator of tissue and bowel perfusion.

The investigators hypothesise that ICG-NIRF is a suitable, reliable and precise method of visualisation of the blood supply and bowel perfusion in the area of ileal pouch formation and the ileal pouch-anal anastomosis.

In this prospective, non-randomized cohort study, restorative proctocolectomy with ileal pouch reconstruction and ileal pouch-anal anastomosis is performed according to standard of care for medically-refractory ulcerative colitis (UC), UC-associated neoplasia, medically-refractory Crohn´s colitis, colorectal carcinoma or familial adenomatous polyposis (FAP) in open or laparoscopic surgery, according to the surgeon's choice.

Written informed consent for participation and ICG-administration is obtained one day before surgery.

Intraoperatively, Indocyanine Green (VerDye, Diagnostic Green GmbH, Aschheim Germany, 25 mg vials) is dissolved in 5 mL sterile water to yield a 5 mg/mL concentration. It will then be administered intravenously at three consecutive time points as a bolus of 2 ml per time point at the most. The overall dose of ICG will amount to no more than 30mg of ICG per patient.

Real-time intraoperative visualization is performed with the SpectrumTM Fluorescence Imaging Platform (Quest Innovations, Middenmeer, The Netherlands) directly after each ICG injection assessing bowel perfusion at three different time points respectively: before and after J-Pouch construction by stapler anastomosis and after ileoanal anastomosis formation.

Clinical data and follow-up Clinical data is be collected from all patients regarding anastomotic leak, bowel ischemia and necrosis as well as 30 day postoperative morbidity, mortality and length and cost of hospital stay.

Subjective data analysis will performed using Microsoft Excel® and IBM SPSS®.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* capability of signing the informed consent
* diagnosis of therapy resistent ulcerative colitis, colorectal cancer, Crohn's disease, familial adenomatous polyposis
* restaurative proctocolectomy (RPC) with reconstruction through ileal pouch formation and ileal pouch-anal anastomosis (IPAA) is possible and medically indicated
* ASA score ≤ 3

Exclusion Criteria:

* coexistent malignant tumor of a different ethology
* liver disfunction (MELD score > 10)
* ICG (indocyanine green) specific exclusion criteria as per literature (intolerance to indocyanine green or sodium iodide, iodine allergy, hyperthyroidism, autonomous thyroid adenoma, focal or diffuse autonomies of the thyroid, previously badly tolerated injection of ICG)
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | 30 days
  occurrence of anastomotic leak within 30 days of surgery

SECONDARY OUTCOMES:
Operative and post-operative complications | 30 days
  Clavien-Dindo for complication-level classification
Length of post-operative hospital stay | 100 days
  length in days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
this will be determinable at a later point when more data is available

REFERENCES:
- [Background] McDermott FD, Heeney A, Kelly ME, Steele RJ, Carlson GL, Winter DC. Systematic review of preoperative, intraoperative and postoperative risk factors for colorectal anastomotic leaks. Br J Surg. 2015 Apr;102(5):462-79. doi: 10.1002/bjs.9697. Epub 2015 Feb 19. PMID 25703524
- [Background] Perbeck L, Lindquist K, Proano E, Liljeqvist L. Correlation between fluorescein flowmetry and laser Doppler flowmetry. A study in the intestine (ileoanal pouch) in man. Scand J Gastroenterol. 1990 May;25(5):520-4. doi: 10.3109/00365529009095524. PMID 2163097
- [Background] Hallbook O, Johansson K, Sjodahl R. Laser Doppler blood flow measurement in rectal resection for carcinoma--comparison between the straight and colonic J pouch reconstruction. Br J Surg. 1996 Mar;83(3):389-92. doi: 10.1002/bjs.1800830330. PMID 8665202
- [Background] van den Bos J, Jongen ACHM, Melenhorst J, Breukink SO, Lenaerts K, Schols RM, Bouvy ND, Stassen LPS. Near-infrared fluorescence image-guidance in anastomotic colorectal cancer surgery and its relation to serum markers of anastomotic leakage: a clinical pilot study. Surg Endosc. 2019 Nov;33(11):3766-3774. doi: 10.1007/s00464-019-06673-6. Epub 2019 Feb 1. PMID 30710314
- [Background] van den Bos J, Al-Taher M, Schols RM, van Kuijk S, Bouvy ND, Stassen LPS. Near-Infrared Fluorescence Imaging for Real-Time Intraoperative Guidance in Anastomotic Colorectal Surgery: A Systematic Review of Literature. J Laparoendosc Adv Surg Tech A. 2018 Feb;28(2):157-167. doi: 10.1089/lap.2017.0231. Epub 2017 Nov 6. PMID 29106320
- [Background] Degett TH, Andersen HS, Gogenur I. Indocyanine green fluorescence angiography for intraoperative assessment of gastrointestinal anastomotic perfusion: a systematic review of clinical trials. Langenbecks Arch Surg. 2016 Sep;401(6):767-75. doi: 10.1007/s00423-016-1400-9. Epub 2016 Mar 11. PMID 26968863